CLINICAL TRIAL: NCT00710749
Title: An Open Prospective Multicenter Study Comparing the Urine Flow Measurements of Standard Clinic Flow Measurements vs Comercially Available Portable Digital Flow Meters and a Disposable Flow Meter in a Crossover and Randomized Order on Male BPH Subjects
Brief Title: The Value of Multiple Urine Flow Rate Measurements in Male Benign Prostatic Hyperplasia (BPH) Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: YA-FLO-0001
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Bladder Outlet Obstruction; Lower Urinary Tract Symptoms
Keywords: Lower urinary tract symptoms leading to lower flow rates
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Disposable device first, then Digital device (Experimental)
  Interventions: Device: Disposable device; Device: Digital device; Device: Clinic flow measurement
- Digital device first, then Disposable device (Experimental)
  Interventions: Device: Disposable device; Device: Digital device; Device: Clinic flow measurement

INTERVENTIONS:
Device: Disposable device — Disposable urine flow meter
Device: Digital device — Digital urine flowmeter
Device: Clinic flow measurement — Clinic gold standard flow measurement

SUMMARY:
Crossover comparison of different flow meters with a digital home flow meter as a reference. Main hypothesis: Reapeated home flow measurements with a disposable device will provide a better understanding of the patients urinary flow than a single measurement performed in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Males aged 45-85 years
* >60% of the voiding volume is above 100 ml per voiding verified by a urinary diary
* Able to read write and understand given instructions

Exclusion Criteria:

* Patients practicing CIC
* Ongoing symptomatic UTI
* Known Neurological Disease that is affecting the bladder function
* Known past or present alcohol or drug abuse
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study site)
* Previous enrolment or randomisation of treatment in the present study.
* Suspected poor compliance based on less than 80 % compliance to voiding diary
* Severe non-compliance to protocol as judged by the investigator and/or Astra Tech
* On alpha-blocker or 5-alpha reductase inhibitor treatment, treatment started less than 2 months prior to enrolment
* Clinic flow below 100 ml

Ages: 45 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Jacobsson, Prof., Study Chair — Dentsply Sirona Implants and Consumables
Locations (4):
- David Geffen school of Medicine at UCLA, Department of Urology, Los Angeles, California, United States
- UMC ST Radboud Nijmegen, Department of Urology, Nijmegen, Netherlands
- Klinika Urology, Akademi Medycznej, Warsaw, Poland
- Clinical Research Unit, Morriston Hospital, Swansea NHS Trust, Swansea, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Disposable Device First, Then Digital Device: 12 voidings recorded with the disposable device in the first intervention period, followed by 12 voidings recorded with the digital device in the second intervention period.
- Digital Device First, Then Disposable Device: 12 voidings recorded with the digital device in the first intervention period, followed by 12 voidings recorded with the disposable device in the second intervention period.
Period: Clinic Baseline Recording
Arm/Group | Disposable Device First, Then Digital Device | Digital Device First, Then Disposable Device
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: First Intervention
Arm/Group | Disposable Device First, Then Digital Device | Digital Device First, Then Disposable Device
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Disposable Device First, Then Digital Device | Digital Device First, Then Disposable Device
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to use the Disposable device first and the Digital device first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 60
Region of Enrollment [Number; unit: participants]
  United States | 2
  Poland | 16
  Netherlands | 13
  United Kingdom | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Urine Flow Rate
Description: Measurements with a disposable device and the current clinic gold standard measurement were compared to test the hypothesis that three repeated measurements with the disposable device was as accurate as one clinic flow measurement. A digital device was used as a reference of the most exact way to evaluate each patient's individual flow.
Time Frame: At every voiding event during approximately one week.
Population: Intention to treat analysis. Number of participants analyzed differs between groups since data was missing mainly due to technical problems.
Measure: Mean (Standard Deviation); unit: ml/s
Groups:
- Disposable Device: Voidings recorded with the disposable device in either first intervention period or second intervention period.
- Clinic: Voidings recorded with the clinic gold standard.
- Digital Device: Voidings recorded with the digital device in either first intervention period or second intervention period.
Arm/Group | Disposable Device | Clinic | Digital Device
Number analyzed (Participants) | 57 | 59 | 52
ml/s | 12 (4) | 13 (7) | 16 (8)
Statistical Analysis 1: Comparison: Disposable Device vs Clinic; Test type: Superiority or Other; p = 0.44, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Clinic vs Digital Device; Test type: Superiority or Other; p = 0.0001, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Disposable Device vs Digital Device; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test

ADVERSE EVENTS:
Arm/Group | Disposable Device | Clinic | Digital Device
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days